CLINICAL TRIAL: NCT02452281
Title: Phase I-II Pilot Study to Evaluate the Immune-mediated Effects of an Autologous Tumor-derived Heat Shock Protein-peptide Complex 96 (HSPPC-96) Combined With Ipilimumab in Patients With Therapeutically Unresectable Stage III or Stage IV Malignant Melanoma
Brief Title: Pilot Study to Evaluate the Effects of a Vaccine (HSPPC-96) Combined With Ipilimumab in Patients With Advanced Melanoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI departure, operational issues
Sponsor: Rabih Said (Other)
Collaborators: Agenus Inc. (Industry)
Responsible Party: Sponsor-Investigator, Rabih Said, Assistant Professor, Department of Internal Medicine, Division of Oncology, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-100-41; HSC-MS-14-0070 (Other: UTHSC-H CPHS (IRB))
Record Dates: First submitted 2015-05-13; First posted 2015-05-22 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Melanoma
Keywords: Therapeutically Unresectable; Stage III or Stage IV; Malignant Melanoma; Advanced Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; vitespin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ipilimumab + HSPPC-96 (Experimental): * Ipilimumab is administered intravenously at a dose of 3 mg/kg one day (a minimum of 12 hours and not more than 48 hours) before HSPPC-96 every 21-25 days for a total of 4 cycles.
  * HSPPC-96 is administered at a dose of 25 μg by intradermal injection always 12 - 48 hours following ipilimumab on a weekly basis for the first 4 weeks and then every 3 weeks always 12 - 48 hours after ipilimumab.
  * Length of Treatment: 4 cycles of ipilimumab and at least 6 cycles of HSPPC-96 up to 12 doses.
  * Booster doses of HSPCC-96 following 6 administrations on subsequent cycles will be administered every 21-23 days according to availability of vaccine.
  Interventions: Drug: ipilimumab; Drug: HSPPC-96

INTERVENTIONS:
Drug: ipilimumab — 3 mg/kg, IV one day (a minimum of 12 hours and not more than 48 hours) before HSPPC-96 every 21-25 days for a total of 4 cycles.
  Other Names: Yervoy ®
Drug: HSPPC-96 — 25 μg by intradermal injection always 12 - 48 hours following ipilimumab on a weekly basis for the first 4 weeks and then every 3 weeks always 12 - 48 hours after ipilimumab; for at least 6 cycles of HSPPC-96 up to 12 doses.
  Other Names: heat shock protein-peptide complex 96; Prophage; Vitespen

SUMMARY:
The purpose of this research study is to see if the combination of HSPPC-96 and ipilimumab is safe and effective in the treatment of advanced melanoma. HSPPC-96 is an investigational vaccine created from tissue from the patient's tumor. The vaccine is designed to capture the cancer's "fingerprint." Injection of the vaccine may cause the patient's immune system to recognize and attack any cells with the specific cancer fingerprint. Ipilimumab is a drug approved by the FDA for the treatment of metastatic melanoma that boosts immune response.

DETAILED DESCRIPTION:
This is a randomized, open label, single-center, phase I-II trial to determine the safety, feasibility and immunogenicity of combination treatment of HSPPC-96 and ipilimumab in patients with therapeutically unresectable Stage III or Stage IV malignant melanoma.

The main purpose of this study is to assess whether the administration of the combination of ipilimumab and HSPPC-96 is safe. The rationale for combining the two treatments resides in their respective roles on the immune system as described below and based on the clinical experience collected so far. HSPPC-96 is able to initiate a tumor specific immune response that ipilimumab could theoretically amplify by blocking a checkpoint that naturally down-regulates T cells.

ELIGIBILITY:
Inclusion Criteria:Pre-surgery Inclusion criteria:

* Signed informed consent
* ≥ 18 years of age
* Stage III or Stage IV melanoma according to TNM staging criteria/AJCC version 7 determined by PET/MRI/CT scan
* ECOG score 0 or 1
* Life expectancy ≥6 months
* Candidate for surgical resection with viable melanoma tissue to ascertain ≥ 7 grams of viable cancer tissue (in aggregate), which is equivalent to a ≥ 2 cm lesion on CT/MRI or clinical examination
* Adequate cardiac function (≤ NYHA class II)
* Adequate bone marrow function, including: absolute granulocyte count (ANC) ≥ 1,500x106/L, absolute lymphocyte count (ALC) ≥ 500/mm3, platelets count ≥100,000 x 106/mm3. Adequate liver function including: serum glutamic oxaloacetic transaminases/aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x the upper limit of institutional normal (IULNs), bilirubin ≤ 1.5 mg/dL or 25 µmol/L (SI units). Adequate renal function: BUN and Serum creatinine of ≤ 1.5 mg/dL or 130 µmol/L (SI units)
* Female subjects of childbearing potential and fertile males must agree to use adequate contraception during the course of the study. Adequate contraception includes condoms with contraceptive foam; oral, implantable or injectable contraceptives; contraceptive patch; intrauterine device; diaphragm with spermicidal gel; or a sexual partner who is surgically sterilized or postmenopausal.

  * Post-surgery Inclusion Criteria (must be completed within 4 weeks of surgery)
* Histologically and clinically confirmed Stage III and/or Stage IV malignant melanoma according to TNM Staging Criteria/AJCC version 7 confirmed by PET/CT scan
* Measurable disease for target lesion clinical and radiological monitoring
* ECOG score 0 or 1
* Adequate cardiac function (≤ NYHA class II)
* Adequate bone marrow function, liver, and renal function
* ≥ 6 doses of vaccine for clinical use

Exclusion Criteria: Pre-Surgery Exclusion Criteria:

* Primary mucosal or primary ocular melanomas
* Other malignancies treated within the last five years, except in situ cervix carcinoma or non-melanoma skin cancer
* Primary or secondary immunodeficiency (including immunosuppressive disease, or systemic use of corticosteroids or other immunosuppressive medications)
* Patients with history of HIV1 and 2, HTLV-1, HBV or active HCV.
* Patients with history of connective tissue disorders
* Prior ipilimumab or melanoma vaccine therapy
* Prior therapy with IL-2
* Prior chemotherapy, small molecule targeted therapy, interferon within 3 months prior to enrollment
* Prior investigational products administration within 4 weeks prior to enrollment
* Prior splenectomy
* Symptomatic CNS metastases or spinal cord compression
* Uncontrolled infection or other serious medical illnesses
* Any medical conditions that, in the opinion of the investigator, would preclude use of ipilimumab, including ipilimumab hypersensitivity
* Women who are pregnant or breast-feeding
* Concurrent participation in investigational trials

  * Post-surgery Exclusion Criteria (must be completed within 4 weeks of surgery):
* Emergence of contraindicated clinical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
All enrolled patients who receive at least one dose of study drug (HSPPC-96) will be evaluated for safety. (adverse events) | 2 years
  AEs will be coded by system organ class and preferred term using MedDRA. AEs will be summarized using descriptive statistics. Descriptive statistics will contain the number and percentage of patients who experience at least 1 AE, AEs related to study treatment, SAEs, SAEs related to study treatment, grade 3, 4 or 5 AEs, and grade 3, 4 or 5 AEs related to study treatment. In addition, the number and percentage of patients who discontinue treatment for any reason, including discontinuation due to an AE, will be provided together with the number and percentage of patients who die.
• To assess immunological response by surrogate markers of immune response and modulation of tumor cellular microenvironment | 2 years
  All enrolled patients who receive at least one full cycle of treatment and have a baseline and at least one post treatment biological specimen available (tissue and/or blood) will be evaluated for immune response.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | tumor evaluations every 12 weeks or until the date of first documented progression or death, whichever came first, assessed up to 24 months
  ORR defined by complete and partial responses.
Progression Free Survival (PFS) | tumor evaluations every 12 weeks or until the date of first documented progression or death, whichever came first, assessed up to 24 months
  Time to recurrence is time from surgery until recurrence or last tumor evaluation without recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Rabih Said, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- UTHealth Memorial Hermann Cancer Center, Houston, Texas, United States